CLINICAL TRIAL: NCT03538587
Title: Feasibility and Preliminary Efficacy of an Enhanced Mindfulness Intervention for Children and Young Adults With High Grade or High-Risk Cancer and Their Caregivers: A Pilot Randomized Controlled Trial
Brief Title: Feasibility and Preliminary Efficacy of a Mindfulness-based Intervention for Children and Young Adults With High Grade or High-Risk Cancer and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Staci Peron, Ph.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 180080; 18-C-0080
Record Dates: First submitted 2018-05-25; First posted 2018-05-29 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Glioblastomas; Sarcoma; Astrocytoma; Brain Cancer; Leukemia
Keywords: Refractory Metastatic Sarcoma; Diffuse Intrinsic Pontine Glioma DIPG; Relapsed-Refractory Leukemia; Meditation; Quality of Life
MeSH Terms: conditions — Glioblastoma; Sarcoma; Astrocytoma; Brain Neoplasms; Leukemia; Diffuse Intrinsic Pontine Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 Enhanced Mindfulness Intervention (EMI) - Immediate Group (Active Comparator): Participate in an in-person session followed by a series of at-home assignments, and two booster sessions.
  Interventions: Behavioral: Enhanced Mindfulness Intervention
- Arm 2 Control Group - Psychoeducation Group (Active Comparator): Participants will briefly meet with a member of the research team who will assess parent and child coping, and provide the child- caregiver dyad educational material about coping with cancer
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Enhanced Mindfulness Intervention — The 8-week EMI will consist of one initial in-person session with the participant and parent, a series of at home assignments, and two "booster" sessions. The psychoeducation group will be given educational material about coping with cancer.
  Arms: Arm 1 Enhanced Mindfulness Intervention (EMI) - Immediate Group
Behavioral: Psychoeducation — The psychoeducation group will be offered the opportunity to participate in the EMI 8 weeks post-baseline.
  Arms: Arm 2 Control Group - Psychoeducation Group

SUMMARY:
Background:

People cope with cancer in different ways. Mindfulness means focusing on the present moment with an open mind. Researchers want to see if this can help children and young adults with a high-grade high-risk cancer with poor prognosis.

Objective:

To learn if mindfulness is feasible and acceptable for children and young people with high-grade high-risk cancer with poor prognosis and their caregivers.

Eligibility:

Children ages 5-24 with a high-grade or high-risk cancer, with a caregiver who agrees to do the study

Must have internet access (participants may borrow an iPod for the study)

Must speak English

Design:

All participants will complete questionnaires. These will be about feelings, physical well-being, quality of life, and mindfulness.

Researchers will review children's medical records.

Participants will be randomly put in the mindfulness group or the standard care group.

Participants in the standard care group will:

Get general recommendations for coping with cancer

Have check-in sessions 1 and 3 weeks after starting. These will last about 10 minutes each.

After participants finish the standard care group, they may be able to enroll in the mindfulness group.

Participants in the mindfulness group will:

Attend an in-person mindfulness training session. The child participant will meet with one research team member for 90 minutes while the parent participant meets with another. Then they will come together for a half hour.

Practice mindfulness exercises at least 4 days a week for 8 weeks.

Be asked to respond to weekly emails or texts asking about their mindfulness practice

Get a mindfulness kit with things to help them do their mindfulness activities at home.

Have a 30-minute check-in with their coach 1 and 3 weeks after starting. This can be in person or by video chat.

All participants (from both groups) will be asked to answer follow-up questions about 8 and 16 weeks after starting the study. Participants will be paid $20 for each set of questionnaires they complete to thank them for their time.

...

DETAILED DESCRIPTION:
Background

* Children and young adults diagnosed with a high-grade or high-risk cancer (e.g., diffuse intrinsic pontine glioma, glioblastoma multiforme, relapsed-refractory leukemia, refractory metastatic sarcomas) face a poor prognosis given limited curative options.
* Recent research has indicated that this population of patients and their parents experience elevated stress and poorer health-related quality of life (HRQL) relative to normative samples.
* Recently published psychosocial standards of care in pediatric oncology strongly recommend that children diagnosed with cancer and their caregivers receive early and continued assessment of their wellbeing and have access to interventions to optimize functioning and HRQL. In addition, there is increasing recognition of the importance of palliative interventions early in the disease trajectory.
* Despite this recommendation, minimal research has examined supportive care interventions for this population early in the disease trajectory.
* Mindfulness-based interventions (MBIs) have empirical support for their feasibility and efficacy in alleviating emotional distress and physical symptoms in children and adults with chronic health conditions, including terminally-ill patients and their caregivers.

Objectives

-To assess the feasibility of an enhanced mindfulness intervention (EMI) in children and young adults (ages 5-24 years) with a high-grade or high-risk cancer with poor prognosis and one of their primary caregivers.

Eligibility

* Children and young adults ages 5-24 years and a parent or adult primary caregiver
* Diagnosis of a high-grade or high-risk cancer with poor prognosis
* English speaking
* Must have access to a mobile device or computer with internet.
* Potential participants will be excluded if there is evidence of pre-morbid severe cognitive or psychiatric disability in parent or child that would impair their capacity for participation, or if there is evidence of clinical disease progression at the time of referral to this study, such that it would prevent the child from engaging in the intervention.

Design

* This is a pilot randomized controlled trial that will compare feasibility and preliminary efficacy of an 8-week enhanced mindfulness intervention (EMI) group (n=10 dyads) compared to a psychoeducation control group (n=10 dyads).
* All participants will complete measures of feasibility (primary outcome) and exploratory outcomes at baseline and following the 8-week intervention. Exploratory measures will include emotional (e.g., depression, anxiety) and physical (e.g., pain, fatigue) wellbeing, as well as baseline mindfulness/self-compassion.
* The 8-week EMI will consist of one initial in-person session with the child and parent, a series of at-home assignments, and two booster sessions. The psychoeducation group will be given educational material about coping with cancer.
* The psychoeducation group will be offered the opportunity to participate in the EMI 8 weeks post-baseline

ELIGIBILITY:
* INCLUSION CRITERIA FOR CHILDREN:
* Patients diagnosed with a high-risk/high-grade cancer (e.g., high-grade brain tumors, relapsed/refractory acute lymphoblastic leukemia, acute myeloid leukemia, high-grade sarcoma) characterized by poor prognosis (e.g., estimated 5-year survival rate <30% based on scientific consensus in the literature, where available, or by expert physician report), as confirmed by medical record review.
* Patients with active disease
* Age greater than or equal to 5 years and less than or equal to 24 years of age
* Must be able to speak and understand English.
* Must have a parent or adult primary caregiver willing to participate in the study.
* Ability of subject or parent/guardian to understand and the willing to sign a written informed consent document.
* Must have access to a computer/mobile device and the internet.

EXCLUSION CRITERIA FOR PATIENTS:

* Patients will be excluded if there is evidence of pre-morbid severe cognitive or psychiatric disability that would impair their capacity for participation or completion of evaluations in the judgment of the investigators.
* Evidence of disease progression at the time of referral to this study to the extent that it would impede participation or completion of evaluations as determined by the medical advisory investigator in conjunction with the study principal investigator (PI)/adjunct PI.
* Patients with treatment-related sequelae so severe that they would be unable to complete the study-related evaluations or intervention (e.g., treatment toxicity) as determined by the medical advisory investigator in conjunction with the study PI/adjunct PI.

INCLUSION CRITERIA FOR PARENT OR ADULT PRIMARY CAREGIVER:

* Must be a parent or primary caregiver of a child (age 5 to 24 years of age) who has been diagnosed with a high-grade/high risk tumor that carries poor prognosis (as defined above); and must live in the same household as the patient for a majority of the time.
* Must have a child willing to participate in the study
* Must be able to speak and understand English.
* Ability of subject to understand and the willing to sign a written informed consent document.
* Must have access to a computer/mobile device and the internet.

Ages: 5 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Staci M Peron, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-C-0080.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 Enhanced Mindfulness Intervention (EMI) - Immediate Group: Arm 1/Enhanced Mindfulness Intervention (EMI) Group - Participate in an in-person session followed by a series of at-home assignments, and two booster sessions.
  Enhanced Mindfulness Intervention: The 8-week EMI will consist of one initial in-person session with the child participant and parent (= 1 dyad), a series of at home assignments, and two "booster" sessions.
- Arm 2 Control Group - Psychoeducation Group: Arm 2 Control Group - Psychoeducation Group Participants will briefly meet with a member of the research team who will assess parent and child coping and provide the child- caregiver dyad educational material about coping with cancer.
  Psychoeducation: The dyads (= 1 child participant and 1 caregiver) in the psychoeducation group will be given educational material about coping with cancer. The psychoeducation group will be offered the opportunity to participate in the EMI 8 weeks post-baseline.
Period: Overall Study
Arm/Group | Arm 1 Enhanced Mindfulness Intervention (EMI) - Immediate Group | Arm 2 Control Group - Psychoeducation Group
Started | 4 (2 dyads (each dyad = 1 child, 1 parent)) | 6 (3 dyads (each dyad = 1 child, 1 parent))
Child Participants | 2 | 3
Parent Participants | 2 | 3
Completed | 2 (1 dyad (each dyad = 1 child, 1 parent)) | 2 (1 dyad (each dyad = 1 child, 1 parent))
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Arm 1 Enhanced Mindfulness Intervention (EMI) - Immediate Group: Arm 1/Enhanced Mindfulness Intervention (EMI) Group - Participate in an in-person session followed by a series of at-home assignments, and two booster sessions.
  Enhanced Mindfulness Intervention: The 8-week EMI will consist of one initial in-person session with the participant and parent, a series of at home assignments, and two "booster" sessions. The psychoeducation group will be given educational material about coping with cancer.
- Arm 2 Control Group - Psychoeducation Group: Arm 2 Control Group - Psychoeducation Group Participants will briefly meet with a member of the research team who will assess parent and child coping and provide the child- caregiver dyad educational material about coping with cancer.
  Psychoeducation: The psychoeducation group will be offered the opportunity to participate in the EMI 8 weeks post-baseline.
- Total: Total of all reporting groups
Arm/Group | Arm 1 Enhanced Mindfulness Intervention (EMI) - Immediate Group | Arm 2 Control Group - Psychoeducation Group | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 3 | 5
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Number of participants analyzed = child and parent participants.
  years
    Child participants: number analyzed (Participants) | 2 | 3 | 5
    Child participants | 11.0 (2.82) | 13.33 (4.73) | 12.16 (3.77)
    Parent participants: number analyzed (Participants) | 2 | 3 | 5
    Parent participants | 44.0 (5.66) | 42.0 (6.56) | 43.0 (6.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 1 | 4 | 5
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 10
School Setting for Child Participants [Count of Participants; unit: Participants] — Population: Analyzed = child participants only.
  Participants
    Public: number analyzed (Participants) | 2 | 3 | 5
    Public | 1 | 3 | 4
    Home School: number analyzed (Participants) | 2 | 3 | 5
    Home School | 1 | 0 | 1
Current School Grade Level for Child Participants [Count of Participants; unit: Participants] — Population: Analyzed = child participants only.
  Participants
    Grade 12: number analyzed (Participants) | 2 | 3 | 5
    Grade 12 | 0 | 1 | 1
    Grade 10: number analyzed (Participants) | 2 | 3 | 5
    Grade 10 | 0 | 1 | 1
    Grade 7: number analyzed (Participants) | 2 | 3 | 5
    Grade 7 | 1 | 0 | 1
    Grade 4: number analyzed (Participants) | 2 | 3 | 5
    Grade 4 | 1 | 0 | 1
    Grade 3: number analyzed (Participants) | 2 | 3 | 5
    Grade 3 | 0 | 1 | 1
Occupation Status for Parent Participants [Count of Participants; unit: Participants] — Population: Analyzed = parent participants only.
  Participants
    Working: number analyzed (Participants) | 2 | 3 | 5
    Working | 1 | 1 | 2
    Not working: number analyzed (Participants) | 2 | 3 | 5
    Not working | 0 | 1 | 1
    On leave: number analyzed (Participants) | 2 | 3 | 5
    On leave | 1 | 0 | 1
    Disability: number analyzed (Participants) | 2 | 3 | 5
    Disability | 0 | 1 | 1
Marital Status [Count of Participants; unit: Participants] — Population: Analyzed = parent participants only.
  Participants
    Single: number analyzed (Participants) | 2 | 3 | 5
    Single | 0 | 1 | 1
    Married: number analyzed (Participants) | 2 | 3 | 5
    Married | 2 | 2 | 4
Number of Parent Participants Working (Hours/Weeks) [Count of Participants; unit: Participants] — Population: Analyzed = parent participants only.
  Participants
    40 Hours/Week: number analyzed (Participants) | 2 | 3 | 5
    40 Hours/Week | 0 | 1 | 1
    37 Hours/Week: number analyzed (Participants) | 2 | 3 | 5
    37 Hours/Week | 1 | 0 | 1
    Not Working: number analyzed (Participants) | 2 | 3 | 5
    Not Working | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eligible Dyads (Parent-child) Who Enroll During a Two-year Period
Description: Percentage of eligible dyads (1 parent, 1 child) who enroll during a two-year period (the number of dyads who enrolled divided by the number of dyads who were found eligible).
Time Frame: 2 years
Population: Each dyad = 1 child, 1 parent. Two dyads were analyzed in group 1 (i.e., 2 children, 2 parents), and three dyads were analyzed in group 2 (i.e., 3 children, 3 parents).
Measure: Number; unit: percentage of dyads
Arm/Group | Arm 1 Enhanced Mindfulness Intervention (EMI) - Immediate Group | Arm 2 Control Group - Psychoeducation Group
Number analyzed (Participants) | 2 | 3
percentage of dyads | 100 | 100

2. Primary Outcome: Percent of Participants (Parent/Child) With Treatment Specific Retention Among All Randomized Participants, With a Target Retention Rate of 70% Over the 8 Week EMI/Control Period
Description: Percent of participants who completed the study among those who enrolled and were randomized, with a target retention rate of 70% over the 8 Week EMI/control period.
Time Frame: 8 weeks from study entry
Measure: Number; unit: percentage of participants(parent/child)
Arm/Group | Arm 1 Enhanced Mindfulness Intervention (EMI) - Immediate Group | Arm 2 Control Group - Psychoeducation Group
Number analyzed (Participants) | 4 | 6
percentage of participants(parent/child) | 50 | 33

3. Primary Outcome: Percent of Participants Who Completed a Mean of 4 Days/Week At-home Practices or More
Description: Compliance with at-home practices (e.g., at home assignments), with a proposed target rate of at least 4 out of 7 days per week on average over the 8 weeks. This will be measured in phone interviews and recorded on a study form.
Time Frame: For 8 weeks from study entry
Measure: Number; unit: percentage of participants
Groups:
- Arm 1 Enhanced Mindfulness Intervention (EMI) - Immediate Group: Arm 1 Enhanced Mindfulness Intervention (EMI) - Immediate Group - Participate in an in-person session followed by a series of at-home assignments, and two booster sessions.
  Enhanced Mindfulness Intervention: The 8-week EMI will consist of one initial in-person session with the participant and parent, a series of at home assignments, and two "booster" sessions. The psychoeducation group will be given educational material about coping with cancer.
Arm/Group | Arm 1 Enhanced Mindfulness Intervention (EMI) - Immediate Group | Arm 2 Control Group - Psychoeducation Group
Number analyzed (Participants) | 4 | 6
percentage of participants | 25 | 0

4. Primary Outcome: Score on a Scale for Caregiver/Children Reports of Satisfaction on the Feasibility Questionnaire
Description: The Feasibility questionnaire is a 12-item measure created by the researchers to assess satisfaction with the study. The first 6 items are on 5-point Likert scales and ask how helpful various aspects of the intervention were. Satisfaction scores are the mean of items 1-6 for both the caregiver and child forms, with possible scores ranging from 1 to 5. Higher scores represent more satisfaction. For youth ages 8+ and caregivers, average item scores of >3.0 reflect adequate satisfaction.
Time Frame: 8 weeks from study entry
Population: Each dyad = 1 child, 1 parent. Half a dyad was analyzed in group 1 (i.e., 1 child), and 1 dyad (i.e., 1 child, 1 parent) was analyzed in group 2. Measure type "Number" is used instead of "Mean" because you cannot compute a mean from only one data point. Unfortunately, not enough participants completed this study measure to calculate means and standard deviations.
Measure: Number; unit: score on a scale
Arm/Group | Arm 1 Enhanced Mindfulness Intervention (EMI) - Immediate Group | Arm 2 Control Group - Psychoeducation Group
Number analyzed (Participants) | 1 | 2
score on a scale
  Child Participants: number analyzed (Participants) | 1 | 1
  Child Participants | 1.83 | 3.5
  Parent Participants: number analyzed (Participants) | 0 | 1
  Parent Participants |  | 3.67

5. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 2-3 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Enhanced Mindfulness Intervention (EMI) - Immediate Group | Arm 2 Control Group - Psychoeducation Group
Number analyzed (Participants) | 4 | 6
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 2-3 months.
Groups:
- Arm 1 Enhanced Mindfulness Intervention (EMI) - Immediate Group: Arm 1 Enhanced Mindfulness Intervention (EMI) - Immediate Group
  Arm 1 Enhanced Mindfulness Intervention (EMI) - Immediate Group - Participate in an in-person session followed by a series of at-home assignments, and two booster sessions.
  Enhanced Mindfulness Intervention: The 8-week EMI will consist of one initial in-person session with the participant and parent, a series of at home assignments, and two "booster" sessions. The psychoeducation group will be given educational material about coping with cancer.
Arm/Group | Arm 1 Enhanced Mindfulness Intervention (EMI) - Immediate Group | Arm 2 Control Group - Psychoeducation Group
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 0/4 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/87/NCT03538587/Prot_SAP_000.pdf
  • Informed Consent Form: Cohort Standard Consent (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/87/NCT03538587/ICF_001.pdf
  • Informed Consent Form: Cohort Assent 12-17 years old (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/87/NCT03538587/ICF_002.pdf
  • Informed Consent Form: Cohort Caregiver Consent (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/87/NCT03538587/ICF_003.pdf